CLINICAL TRIAL: NCT05141760
Title: Assessing 18F-PSMA-1007 Positron Emission Tomography and Magnetic Resonance Imaging in the Primary Staging of Prostate Cancer Patients
Brief Title: 18F-PSMA PET and MRI in the Primary Staging of Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Urological Association Scholarship Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREBA.CC-21-0073
Record Dates: First submitted 2021-11-09; First posted 2021-12-02 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PSMA-1007 Positron Emission Tomography (PET) scan and 3T Magnetic Resonance Imaging (MRI) — Additional staging PET and MRI scan prior to prostatectomy and lymph node dissection

SUMMARY:
This prospective phase II study assesses the accuracy of second generation prostate specific membrane antigen (PSMA) positron emission tomography (PET; utilizing 18F-PSMA-1007)) and multiparametric magnetic resonance imaging (MRI) for locoregional staging of clinically significant prostate cancer in men undergoing radical prostatectomy and bilateral pelvic lymph node dissection. The design will be a multicenter validating-paired cohort study using radical prostatectomy and pelvic lymph node dissection as the gold standard comparator. Each patient will undergo both 18F-PSMA-1007 PET and 3T MRI allowing comparison of each imaging modality within each subject. Furthermore, PET and MRI will be compared to standard-of-care imaging techniques (CT abdomen/pelvis and 99mTc-MDP Bone scan).

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal medical decision makers will sign an informed consent prior to entering the study.
2. Adult patient (≥ 18 years old) with a diagnosis of at least Gleason Grade Group 2 prostate cancer.
3. Appropriate staging investigations have been performed prior to the participation in the study (i.e. CT abdomen/pelvis and 99mTc-MDP bone scan)

Exclusion Criteria:

1. Unable to obtain consent
2. Weight >250 kg (weight limitation of scanners)
3. Unable to lie flat for 30 minutes to complete the PET or MRI imaging
4. Severe claustrophobia precluding image acquisition
5. Lack of intravenous access
6. Non-MRI compatible pacemaker or hardware
7. eGFR < 40 mL/min/1.73 m2 and/or a history of a severe reaction to MRI contrast
8. Prior androgen deprivation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Tumor T-staging | Through study completion, this is expected to be reviewed within 1 year of imaging
  Differentiate Unilateral vs. Bilateral Tumor (i.e. T2a vs. T2b), Identify extracapsular extension (T3a) or Seminal vesicle invasion (T3b)

SECONDARY OUTCOMES:
Sensitivity of PSMA-1007 PET | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against PSMA-1007 PET
Sensitivity of MRI | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against MR imaging
Specificity of PSMA-1007 PET | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against PSMA-1007 PET
Specificity of MRI | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against MR imaging
Negative Predictive Value of PSMA-1007 PET | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against PSMA-1007 PET
Negative Predictive Value of MRI | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against MR imaging
Positive Predictive Value of PSMA-1007 PET | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against PSMA-1007 PET
Positive Predictive Value of MRI | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against MRI
Nodal Staging | Through study completion, this is expected to be reviewed within 1 year of imaging
  Accuracy of nodal disease on PSMA-1007 PET and MRI compared to bone scan + CT
Metastatic Staging | Through study completion, this is expected to be reviewed within 1 year of imaging
  Accuracy of PSMA-1007 PET and MRI compared to bone scan + CT
Longest Tumor diameter | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare final histology against PSMA-1007 PET and MRI measurements
Identification of dominant lesion | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare rate of dominant lesion identification of PSMA-1007 PET and MRI against final histology
Identification of non-dominant lesion | Through study completion, this is expected to be reviewed within 1 year of imaging
  Compare rate of non-dominant lesion identification of PSMA-1007 PET and MRI against final histology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No